CLINICAL TRIAL: NCT01989585
Title: Phase I/II Study of Dabrafenib, Trametinib, and Navitoclax in BRAF Mutant Melanoma (Phase I and II) and Other Solid Tumors (Phase I Only)
Brief Title: Testing the Addition of Navitoclax to the Combination of Dabrafenib and Trametinib in People Who Have BRAF Mutant Melanoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02103; NCI-2013-02103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-424; 18-716; 9466 (Other: Dana-Farber - Harvard Cancer Center LAO); 9466 (Other: CTEP); U01CA062490 (NIH); U01CA132194 (NIH); UM1CA186688 (NIH); UM1CA186709 (NIH); UM1CA186716 (NIH); NCT01970956 (obsolete NCT alias)
Record Dates: First submitted 2013-11-18; First posted 2013-11-21 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Malignant Solid Neoplasm; Metastatic Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Biopsy; Specimen Handling; dabrafenib; Magnetic Resonance Spectroscopy; navitoclax; trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (dabrafenib, trametinib) (Experimental): ARM I: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, MRI or CT, biopsy, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Other: Pharmacological Study; Drug: Trametinib
- Arm II (dabrafenib, trametinib, and navitoclax) (Experimental): Patients receive navitoclax PO QD days -7 to -1 of cycle 1 only. Patients also receive dabrafenib PO BID, trametinib PO QD, and navitoclax PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, MRI or CT, biopsy, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib; Procedure: Echocardiography Test; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Navitoclax; Other: Pharmacological Study; Drug: Trametinib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK 2118436; GSK 2118436A; GSK-2118436; GSK-2118436A; GSK2118436; GSK2118436A
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo multigated acquisition scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Navitoclax — Given PO
  Other Names: A-855071.0; ABT-263; BcI-2 Family Protein Inhibitor ABT-263
  Arms: Arm II (dabrafenib, trametinib, and navitoclax)
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase I/II trial studies the side effects and best dose of dabrafenib, trametinib, and navitoclax and to see how well they work in treating patients with BRAF mutant melanoma or solid tumors that has spread from where it first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Navitoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of tumor cells by blocking Bcl-2, a protein needed for tumor cell survival. Giving navitoclax, dabrafenib, and trametinib may help shrink tumors in patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD), toxicity, and safety profile of navitoclax when given in combination with dabrafenib and trametinib in patients with BRAF-mutant solid tumors. (Phase I) II. To estimate the complete response (CR) rate in patients with BRAF-mutant melanoma treated with dabrafenib, trametinib, and navitoclax as compared to the historical control dabrafenib and trametinib combination (DT). (Phase II) III. To compare the maximal tumor regression in patients with BRAF-mutant melanoma treated with dabrafenib, trametinib versus dabrafenib, trametinib, and navitoclax. (Phase II)

SECONDARY OBJECTIVES:

I. To describe pharmacodynamics effects of treatment with dabrafenib, trametinib, and navitoclax on both serial tumor biopsies and serial blood draws in a small subset of patients treated with BRAF-mutant melanoma. (Phase I) II. To describe the pharmacokinetics of treatment with dabrafenib, trametinib, and navitoclax. (Phase I) III. To compare the progression-free survival (PFS), overall survival (OS), and overall response rate (ORR) in patients with BRAF-mutant melanoma treated with dabrafenib, trametinib, versus dabrafenib, trametinib, and navitoclax. (Phase II) IV. To compare the degree of apoptosis induced in on-treatment biopsies of patients with BRAF-mutant melanoma treated with dabrafenib, trametinib versus dabrafenib, trametinib, and navitoclax. (Phase II) V. To explore other pharmacodynamic effects in on-treatment biopsies of patients with BRAF-mutant melanoma treated with either dabrafenib, trametinib versus dabrafenib, trametinib, and navitoclax including cell proliferation (Ki-67), proteomics (reverse-phase protein microarrays [RPPA]), and B-cell chronic lymphocytic leukemia (CLL)/lymphoma 2 (BCL-2) family gene expression analysis. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of dabrafenib, trametinib, and navitoclax followed by a randomized phase II study.

PHASE I: Patients receive navitoclax orally (PO) once daily (QD) on days -7 to -1 of cycle 1 only. Patients also receive dabrafenib PO twice daily (BID), trametinib PO QD, and navitoclax PO QD days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo electrocardiography (ECHO) or multigated acquisition scan (MUGA), magnetic resonance imaging (MRI) or computed tomography (CT), also undergo biopsy, and collection of blood samples throughout the trial.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, MRI or CT, biopsy, and collection of blood samples throughout the trial.

ARM II: Patients receive navitoclax PO QD days -7 to -1 of cycle 1 only. Patients also receive dabrafenib PO BID, trametinib PO QD, and navitoclax PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, MRI or CT, biopsy, and collection of blood samples throughout the trial.

After the completion of study treatment, patients are followed up for clinical evaluation at 28 days and every 3 months thereafter until disease progression or death, whichever comes first. For survival follow up, patients are followed every 12 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I SUBJECTS ONLY: Prior therapy is allowed; for patients enrolled in the Phase I portion of the study, patients may have received any number of prior lines of therapy including treatment with a BRAF and/or MEK inhibitor; prior navitoclax use will not be allowed, unless the patient received < 7 days of navitoclax lead-in on this or another study and had to stop for reasons other than toxicity or disease progression
* Patients must have histologically confirmed, BRAF-mutant (V600E/K) melanoma (molecularly confirmed using validated, commercially available assay performed in a Clinical Laboratory Improvement Act [CLIA]-approved laboratory) that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective

  * If test at CLIA-certified lab used a non-Food and Drug Administration (FDA) approved method, information about the assay must be provided; (FDA approved tests for BRAF V600 mutations in melanoma include: THxID BRAF Detection Kit and Cobas 4800 BRAF V600 Mutation Test)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan, MRI, or calipers by clinical exam
* Prior therapy is allowed; for patients enrolled in the Phase II portion of the study, patients may have received prior immunotherapy (including high-dose IL-2, ipilimumab, nivolumab, and other anti-PD1/PDL1 antibodies) or chemotherapy; however prior navitoclax, BRAF inhibitor and/or MEK inhibitor therapy will not be allowed
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of navitoclax in combination with dabrafenib and trametinib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1 x 10^9/L
* Hemoglobin >= 9 g/dl (patients may be transfused to this level)
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal OR > 1.5 x institutional upper limit of normal allowed if direct bilirubin is within normal range
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.3 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 mg/dL OR creatinine clearance >= 50 mL/min/1.73 m^2
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by ECHO
* Patients must have a corrected QT (QTc) interval of less than 480 msec
* The effects of navitoclax, dabrafenib, and trametinib on the developing human fetus are unknown; for this reason, women of child-bearing potential and men with partners of childbearing potential must agree to use adequate contraception (barrier method of birth control, or abstinence; hormonal contraception is not allowed due to drug-drug interactions which can render hormonal contraceptives ineffective) prior to study entry, for the duration of study participation, and for 4 months after completion of study drug administration; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; based on studies in animals, it is also known that dabrafenib may cause damage to the tissue that makes sperm; this may cause sperm to be abnormal in shape and size and could lead to infertility, which may be irreversible; safety and efficacy of the combination of dabrafenib and trametinib in pediatric populations have not been investigated; dabrafenib or trametinib-dabrafenib combination should not be administered to pediatric populations outside clinical trials
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Ability to understand and the willingness to sign a written informed consent document; if a patient has impaired decision-making capacity, a legally authorized representative, patients will be allowed to participate

Exclusion Criteria:

* PHASE I SUBJECTS ONLY: Patients must not have received prior navitoclax, unless the patient received < 7 days of navitoclax lead-in on this or another study and had to stop for reasons other than toxicity or disease progression
* Patients who have had immunotherapy, chemotherapy or radiotherapy within 14 days prior to the first dose of navitoclax, or prior systemic anti-cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or vaccine therapy) within the last 3 weeks prior to first dose of dabrafenib and/or trametinib; chemotherapy regimens without delayed toxicity within the last 2 weeks preceding the first dose of study treatment; biologics will not be allowed within 30 days prior to, or during, navitoclax administration
* Prior navitoclax, BRAF inhibitor, and MEK inhibitor is prohibited; (exceptions for Phase I are described above)
* Patients who are receiving any other investigational agents have received any other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study treatment and during the study
* Patients with treated leptomeningeal or brain metastasis are not eligible unless there is demonstrated stability (documented by imaging) for >= 3 months from any prior treatment of leptomeningeal or brain metastasis. Treatment may include surgery, radiation or systemic therapy. Patients with untreated leptomeningeal or brain metastasis or requiring corticosteroids are not eligible. Subjects on a stable dose of corticosteroids > 1 month or who have been off of corticosteroids for at least 2 weeks can be enrolled with approval of the Cancer Therapy Evaluation Program (CTEP) medical monitor. Subjects must also be off of enzyme-inducing anticonvulsants for > 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to navitoclax, dabrafenib, or trametinib, or excipients or to dimethyl sulfoxide (DMSO)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because navitoclax, dabrafenib, and trametinib may have teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued if the mother is treated with the study drugs
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy that predict to interact with any of the study drugs are ineligible because of the potential for pharmacokinetic interactions with the study drugs; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated; it is not necessary to conduct HIV testing at screening; patients who are HIV-positive with undetectable viral loads, not on interacting antiretroviral therapy, and have CD4 counts above 300/mm^3 may be eligible after discussion with the principal investigator
* History of another malignancy; exception: patients who have been disease-free for 3 years (depending upon tumor type studied or clinical setting, 3 or 5 years can be used; e.g., for advanced melanoma and pancreatic studies 3 years is more appropriate due to aggressiveness of the disease, while 5 years can be more appropriate for prostate or ovarian cancer or adjuvant setting when life expectancy is longer), or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the CTEP medical monitor if unsure whether second malignancies meet the requirements specified above; exception: patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study; prospective RAS testing is not required; however, if the results of previous RAS testing are known, they must be used in assessing eligibility
* History of interstitial lung disease or pneumonitis
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

  * History of RVO or CSR, or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
  * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure > 21 mmHg
* History or evidence of cardiovascular risk including any of the following:

  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec on screening electrocardiography (ECG)
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Abnormal cardiac valve morphology (>= grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study); subjects with moderate valvular thickening should not be entered on study
* Known history of hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); it is not necessary to conduct HBV and HCV testing at screening
* Subject has an underlying condition predisposing them to bleeding or currently exhibits signs of clinically significant bleeding
* Subject has a recent history of non-chemotherapy-induced thrombocytopenic-associated bleeding within 1 year prior to the first dose of study drug
* A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v. 5.0) grade 2 or higher from previous anti-cancer therapy, except alopecia or an endocrine toxicity related to immunotherapy (e.g. thyroiditis/hypothyroidism, adrenal insufficiency, hypophysitis) requiring replacement therapy, at the time of randomization
* Due to the expected dose-limiting toxicity of thrombocytopenia, the following concomitant medications are not allowed during navitoclax administration: clopidogrel, ibuprofen, tirofiban, warfarin, and other anticoagulants, drugs, or herbal supplements that affect platelet function are excluded, with the exception of low-dose anticoagulation medications (such as heparin) that are used to maintain the patency of a central intravenous catheter; aspirin will not be allowed within 7 days prior to the first dose of navitoclax or during navitoclax administration; however, subjects who have previously received aspirin therapy for thrombosis prevention may resume a low dose (i.e., maximum 100 mg QD) of aspirin if platelet counts are stable (>= 50,000/mm^3) through 6 weeks of navitoclax administration; all decisions regarding treatment with aspirin therapy will be determined by the investigator in conjunction with the medical monitor
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
  * Anticoagulants and antiplatelet agents are excluded except for low-dose, aspirin
* Preclinical studies indicate that navitoclax is metabolized by CYP3A4, is a moderate inhibitor of CYP2C8, and is a strong inhibitor of CYP2C9; there is also evidence of interactions with dabrafenib; therefore, caution should be exercised when dosing navitoclax concurrently with CYP2C8 and CYP2C9 substrates; common CYP2C8 substrates include paclitaxel, statins, and glitazones, whereas CYP2C9 substrates include phenytoin; when possible, investigators should switch to alternative medications or monitor the patients closely; CYP3A inhibitors such as ketoconazole and clarithromycin are not allowed 7 days prior to the first dose of navitoclax or during navitoclax administration
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible; current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of permeability-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded; below are a few examples of the agents:

  * Strong inducers of CYP3A or CYP2C8, since concentrations of dabrafenib may be decreased:

    * Antibiotics: rifamycin class agents (e.g., rifampin, rifabutin, rifapentine)
    * Anticonvulsants: carbamazepine, oxcarbazepine, phenobarbital, phenytoin, s-mephenytoin
    * Miscellaneous: bosentan, St. John's wort
  * Strong inhibitors of CYP3A or CYP2C8 since concentrations of dabrafenib may be increased:

    * Antibiotics: clarithromycin, telithromycin, troleandomycin
    * Antidepressants: nefazodone
    * Antifungals: itraconazole, ketoconazole, posaconazole, voriconazole
    * Hyperlipidemia: gemfibrozil
    * Antiretroviral: ritonavir, saquinavir, atazanavir
    * Miscellaneous: conivaptan
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-03-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of the combination of dabrafenib, trametinib, and navitoclax (Phase I) | Up to 28 days
  Determined by dose-limiting toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events.
Proportion of patients with a complete response (CR) (Phase II) | Up to 4 weeks after last study treatment
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, in the cohort of patients treated with dabrafenib, trametinib, and navitoclax (DTN). The proportion of patients with a best response of CR will be presented with a 95% confidence interval calculated using the method of Atkinson and Brown.
Maximal degree of tumor regression (Phase II) | Up to 4 weeks after last study treatment
  A comparison between the maximal tumor regression for patients treated with DTN and dabrafenib and trametinib (DT) will be conducted using a Wilcoxon rank-sum test.

SECONDARY OUTCOMES:
Progression free survival (PFS) (Phase II) | Time from start of treatment to time of progression or death, whichever occurs first, assessed for up to 10 years
  PFS will be summarized using the Kaplan-Meier. Log-rank tests will be used to assess for indications of differences between the two treatment modalities.
Overall survival (OS) (Phase II) | Up to 10 years
  OS will be summarized using the Kaplan-Meier. Log-rank tests will be used to assess for indications of differences between the two treatment modalities.
Objective response rate (ORR) (Phase II) | Up to 4 weeks after last study treatment
  ORRs will be presented with 95% exact, binomial confidence intervals.

OTHER OUTCOMES:
Change in terminal deoxynucleotidyl transferase 2´-deoxyuridine, 5´-triphosphate (dUTP) nick end labeling assay (TUNEL) staining | Baseline to up to 1 week
  Fold changes of TUNEL will be calculated (post/pre). A Wilcoxon rank-sum test will be used to compare the ratios (or equivalently, the difference in the natural logs) of baseline and follow-up levels of TUNEL between DTN and DT treatment arms.
Change in B-cell chronic lymphocytic leukemia/lymphoma 2 (BCL-2) | Baseline to up to 1 week
  Will be primarily descriptive.
Change in Ki67 | Baseline to up to 1 week
  Will be primarily descriptive.
Change in phosphatase and tensin homolog (PTEN) status | Baseline to up to 1 week
  Will be primarily descriptive.
Fold changes in BRAF-mutation assay | Baseline to up to 4 weeks after last study treatment
  Fold-changes in assay response will be calculated (post/pre). Fold changes in the assay will be compared across RECIST responses using the Kruskal-Wallis test. In addition, for assay-based response or progression, the proportions of patients with CR/partial response (PR), stable disease (SD), or progressive disease (PD) will be presented with exact 90% confidence intervals. Assay performance data will be compared with response. The proportions will be summarized and compared using exact confidence intervals. Behavior of the blood assay will be summarized graphically.
Fold changes in tumor burden | Baseline to up to 4 weeks after last study treatment
  Assay fold changes will be compared with fold changes in tumor burden (post/pre). The relationship will be summarized graphically and using the Spearman rank correlation. Differences in the behavior of the assay will be explored using a general linear model of log (fold-change) with study, baseline tumor burden, and log (fold-change tumor burden) as predictors.
Pharmacokinetic parameters, including maximal plasma or serum concentration (Cmax), area under the curve to the last collection point (AUClast), area under the curve for dose interval (AUC0-t), and time of maximal concentration (Tmax) | Pre-treatment, 1, 2, 4, 6, 8, and 24 hours post-treatment on days 1 and 15 of cycle 1, and day 1 of cycles 2, 4, 8, and 12 (each cycle = 28 days)
  Descriptive statistics including mean, standard deviation, coefficient of variation, geometric mean, median, minimum and maximum will be computed for each pharmacokinetic variable; descriptive statistics for natural-log transformed pharmacokinetic variables will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Sullivan, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (49):
- United States (49):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas